CLINICAL TRIAL: NCT00000323
Title: Therapeutic Potential of Kappa-Opioids Against Cocaine
Brief Title: Therapeutic Potential of Kappa-Opioids Against Cocaine - 1
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Other Study IDs: NIDA-10753-1; R01-10753-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2004-05

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders

SUMMARY:
The purpose of this study is to characterize the effects of enadoline compared to hydromorphone and butorphanol.

ELIGIBILITY:
Inclusion Criteria:

opiate experienced, healthy

Exclusion Criteria:

physical dependence on opioids, barbiturates or alcohol

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 1996-07; Study Completion 1998-12

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Walsh, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (BPRU) Bayview Campus, Baltimore, Maryland, United States

REFERENCES:
- [Background] Walsh SL, Strain EC, Abreu ME, Bigelow GE. Enadoline, a selective kappa opioid agonist: comparison with butorphanol and hydromorphone in humans. Psychopharmacology (Berl). 2001 Sep;157(2):151-62. doi: 10.1007/s002130100788. PMID 11594439